CLINICAL TRIAL: NCT05869383
Title: Effect Of Ophiochepalus Striatus Extract On Serum IGF-1 And IL-6 Levels In Elderly Patients With Sarcopenia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universitas Sriwijaya (Other)
Responsible Party: Principal Investigator, Nur Riviati, Head of Geriatric Division RSUP Dr. Mohammad Hoesin Palembang, Principal Investigator, Universitas Sriwijaya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D.XVIII.6.11/ETIK/36/2023
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Results first posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Sarcopenia; Geriatric; Muscle Mass; Muscle Strength; Physical Performance
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Both participant and investigator dont know the intervention that have been given.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Control group get placebo 2x5 grams a day for 14 days
  Interventions: Drug: Placebo
- Ophiochepalus striatus extract (Experimental): Intervention group get Ophiochepalus striatus extract 2x5 grams a day for 14 days
  Interventions: Drug: Ophiochepalus striatus extract

INTERVENTIONS:
Drug: Ophiochepalus striatus extract — Ophiochepalus striatus extract 2x5 grams
  Other Names: VipAlbumin
  Arms: Ophiochepalus striatus extract
Drug: Placebo — Placebo 2x5 grams
  Other Names: Placebo contain maltodextrin
  Arms: Placebo

SUMMARY:
The goal of this Clinical Trial is to analyze effect of Ophiochepalus striatus extract on serum IGF-1 and IL-6 levels in elderly patients with sarcopenia. The main questions it aims to answer are:

1. Can giving Ophiocephalus striatus extract at a dose of 2x5 grams for 2 weeks increase IGF-1 levels in elderly people with sarcopenia?
2. Can administration of 2x5 grams dose of Ophiocephalus striatus extract for 2 weeks reduce IL-6 levels in elderly with sarcopenia?
3. Can the administration of Ophiocephalus striatus extract at a dose of 2x5 grams for 2 weeks reduce the SARC-F score in elderly people with sarcopenia?
4. Can the administration of Ophiocephalus striatus extract at a dose of 2x5 grams for 2 weeks increase muscle mass in elderly people with sarcopenia?
5. Can the administration of Ophiocephalus striatus extract at a dose of 2x5 grams for 2 weeks increase muscle strength in elderly people with sarcopenia?
6. Can administration of Ophiocephalus striatus extract at a dose of 2x5 grams for 2 weeks improve physical performance in elderly with sarcopenia?

Participants will:

1. Consume Ophiochepalus striatus extract 2x5 grams a day.
2. Checked blood before and after the intervention.
3. Measured muscle mass, muscle strength, and physical performance before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients with sarcopenia diagnosed using AWGS criteria consist of low muscle mass: using the BIA examination tool where men: <7.0kg/m2, women: <5.7kg/m2 plus low muscle strength using a handgrip dynamometer, men: <28kg , female : <18kg or low physical performance using the 6 meter walk test; <1 meter/second.

Exclusion Criteria:

* Chronic liver disease (cirrhosis of the liver) or severe liver dysfunction or increased SGPT> 3 times the upper limit of normal value
* Impaired kidney function with a glomerular filtration rate <30 ml/minute without hemodialysis
* Acute phase of illness (eg infection, acute arthritis, acute stroke, trauma)
* Malignancy
* Depression according to the geriatric depression scale (Geriatric Depression Scale score> 10)
* History of hypersensitivity to Ophiocephalus striatus
* Refuse to participate in research

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nur Riviati, Principal Investigator — Mohammad Hoesin General Hospital
Locations (1):
- Mohammad Hoesin Central General Hospital, Palembang, South Sumatera, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Riviati N, Legiran L, Saleh I, Indrajaya T, Ali Z, Irfannuddin, Probosuseno. Ophiocephalus striatus Extract Supplementation Decreases Serum IL-6 Levels in Older People with Sarcopenia-A Single-Center Experience. Geriatrics (Basel). 2024 Mar 7;9(2):35. doi: 10.3390/geriatrics9020035. PMID 38525752

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Ophiochepalus Striatus Extract
Started | 40 | 40
Completed | 38 | 40
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ophiochepalus Striatus Extract | Total
Number analyzed (Participants) | 38 | 40 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 9 | 20
  >=65 years | 27 | 31 | 58
Age, Continuous [Median (Full Range); unit: years] | 71 [60 to 88] | 70 [62 to 85] | 71 [60 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 25 | 47
  Male | 16 | 15 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 38 | 40 | 78
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Indonesia | 38 | 40 | 78

OUTCOME MEASURES:

1. Primary Outcome: IGF-1 Levels
Description: IGF-1 serum levels were measured using Cloud-Clone Corp® ELISA reagent with serial numbers 6854322BA3.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: ng/dl
Arm/Group | Placebo | Ophiochepalus Striatus Extract
Number analyzed (Participants) | 38 | 40
ng/dl | 78.92 (21.7) | 77.08 (20.9)

2. Primary Outcome: IL-6 Levels
Description: IL-6 serum levels were measured using Cloud-Clone Corp® ELISA reagent with serial numbers 41148D2B69.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: pg/dl
Arm/Group | Placebo | Ophiochepalus Striatus Extract
Number analyzed (Participants) | 38 | 40
pg/dl | 36.47 (17.45) | 44.51 (23.57)

ADVERSE EVENTS:
Time Frame: 14 days follow up during intervention period
Description: 1. Serious Adverse Events: death, a life-threatening adverse event, and inpatient hospitalization. Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment.
  2. Other Adverse Events: Adverse events that are not Serious Adverse Events.
Arm/Group | Placebo | Ophiochepalus Striatus Extract
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/40
Other Adverse Events (participants affected / at risk) | 6/38 | 8/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=38) | Ophiochepalus Striatus Extract (N=40)
Subjective complaint (Gastrointestinal disorders) | 4 (4) | 6 (6) — Nausea
Subjective complaint (Gastrointestinal disorders) | 2 (2) | 2 (2) — Vomiting

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT05869383/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT05869383/ICF_001.pdf